CLINICAL TRIAL: NCT02735915
Title: Long Term Immunogenicity and Safety Study of GSK Biologicals' Herpes Zoster Subunit (HZ/su) Vaccine 1437173A and Assessment of Re-vaccination With 2 Additional Doses, in Healthy Subjects Aged 60 Years of Age and Older
Brief Title: Study to Evaluate Immunogenicity and Safety of GSK Biologicals' Herpes Zoster Subunit (HZ/su) Vaccine at 9 and 10 Years After Vaccine Administration and Assessment of Re-vaccination With 2 Additional Doses at 10 Years After Initial Vaccination, in Healthy Subjects Aged 60 Years of Age(YOA) and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 204926; 2015-004400-30 (EudraCT Number)
Record Dates: First submitted 2016-04-07; First posted 2016-04-13 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Herpes Zoster
Keywords: Immunogenicity; Safety; Long term follow-up; Adults; Herpes zoster
MeSH Terms: conditions — Herpes Zoster

ARMS (1):
- GSK1437173A vaccine Group (Experimental): Subjects who completed vaccination course of 2 doses of HZ/su vaccine (group 50 μg gE/AS01B) in the study Zoster-003 (NCT00434577) were included in this study. 62 of these subjects further received 1 or 2 additional doses of HZ/su vaccine in the revaccination phase of this study
  Interventions: Biological: Herpes Zoster Vaccine GSK1437173A

INTERVENTIONS:
Biological: Herpes Zoster Vaccine GSK1437173A — Intramuscular injection
  Other Names: HZ/su

SUMMARY:
The purpose of this study is to evaluate the persistence of immune response to the HZ vaccine as well as safety up to 10 years after the first dose of initial vaccination course. This study will also assess immune responses after re-vaccination with 2 additional doses of the HZ/su administered at ten years after first dose of initial vaccination course from study Zoster-003 (NCT00434577).

DETAILED DESCRIPTION:
In this LTFU study (ZOSTER-060), subjects who received 2 doses of HZ/su in the earlier Zoster-003 (NCT00434577) study will be followed up at Month 108/Year 9 and Month 120/Year 10 post first dose of vaccine for safety and immunogenicity (humoral and cellular). In order to assess the effect of re-vaccination with 2 additional doses of HZ/su vaccine, all the subjects will receive 2 additional doses of the HZ/su vaccine, on a 0, 2-month schedule at ten years after the initial vaccination course in study Zoster-003 (NCT00434577), and will be followed for reactogenicity, safety and humoral and cellular immunogenicity (including persistence).

In alignment with the previous persistence timepoints, this study has no control group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits, ability to have scheduled contacts to allow evaluation during the study). Or subjects with a caregiver who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the diary cards, vaccination visits, availability for follow-up contacts).
* Written informed consent obtained from the subject prior to performance of any study specific procedure.
* Previous participation in study ZOSTER-003 (NCT00434577), in group 50 µg gE / AS01B, and who completed the vaccination course (2 doses of HZ/su) in study ZOSTER-003 (NCT00434577).
* Subjects are expected to enter the study (or complete Visit 1) as of the time they turn 108 months after first vaccination of previous vaccination course with HZ/su and not later than 111 months.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine during the period starting 30 days before the first study visit (Day -29 to Day 0), or planned use during the study period.
* Use or anticipated use of immunosuppressants or immune-modifying drugs during the period starting six months prior to study start and during the whole study period. This includes chronic administration of corticosteroids (>14 consecutive days of prednisone at a dose of ≥20 mg/day [or equivalent]), long-acting immune-modifying agents (e.g., infliximab) or immunosuppressive/cytotoxic therapy (e.g., medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders).
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., malignancy, human immunodeficiency virus [HIV] infection).
* Administration or planned administration of a live vaccine in the period starting 30 days before the first dose of study vaccine and ending 30 days after the last dose of study vaccine, or, administration or planned administration of a non-replicating vaccine* within 8 days prior to or within 14 days after either dose of study vaccine.

E.g., inactivated and subunit vaccines, including inactivated and subunit influenza vaccines and pneumococcal conjugate vaccines.

* Previous vaccination against HZ since initial vaccination in Zoster-003.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the study start, or planned administration during the study period.
* History of previous HZ.

Min Age: 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- GSK Investigational Site, Hradec Králové, Czechia
- Germany (4):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
- Sweden (2):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Schwarz TF, Volpe S, Catteau G, Chlibek R, David MP, Richardus JH, Lal H, Oostvogels L, Pauksens K, Ravault S, Rombo L, Sonder G, Smetana J, Heineman T, Bastidas A. Persistence of immune response to an adjuvanted varicella-zoster virus subunit vaccine for up to year nine in older adults. Hum Vaccin Immunother. 2018 Jun 3;14(6):1370-1377. doi: 10.1080/21645515.2018.1442162. Epub 2018 Mar 21. PMID 29461919
- [Background] Hastie A, Catteau G, Enemuo A, Mrkvan T, Salaun B, Volpe S, Smetana J, Rombo L, Schwarz T, Pauksens K, Herve C, Bastidas A, Schuind A. Immunogenicity of the Adjuvanted Recombinant Zoster Vaccine: Persistence and Anamnestic Response to Additional Doses Administered 10 Years After Primary Vaccination. J Infect Dis. 2021 Dec 15;224(12):2025-2034. doi: 10.1093/infdis/jiaa300. PMID 32502272
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who participated in the parent study Zoster-003 (NCT00434577),in GSK1437173A _MD Group and received a complete vaccination course(2 doses of 50 µg GSK1437173A) were offered participation in this Long Term Follow-Up study. A total of 70 subjects met the eligibility criteria & consented to participate in Germany, Sweden and Czech Republic
Pre-assignment Details: Out of 70 subjects originally enrolled (Total enrolled cohort for persistence phase) into the study, 8 subjects were eliminated as subject number was allocated without vaccine administration. Only 62 subjects were vaccinated with at least one dose, forming the Total vaccinated cohort(TVc) for re-vaccination phase.
Groups:
- GSK1437173A Vaccine Group: Subjects who completed vaccination course of 2 doses of HZ/su vaccine (group 50 µg gE/AS01B) in the study Zoster-003 (NCT00434577) were included in this study. 62 of these subjects further received 1 or 2 additional doses of HZ/su vaccine in the revaccination phase of this study
Period: Overall Study
Arm/Group | GSK1437173A Vaccine Group
Started (Started=Number of subjects enrolled into the study (Total enrolled cohort for persistence phase)) | 70
Vaccinated (Vaccinated=Number of subjects that started the Total Vaccinated Cohort (TVc) for revaccination phase) | 62
Completed | 59
Not Completed | 11
Not completed — Not vaccinated but subject ID assigned | 8
Not completed — Withdrawal following SAE | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.3 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Caucasian/European Heritage | 70

OUTCOME MEASURES:

1. Primary Outcome: Anti-glycoprotein (gE) Specific Antibody (Ab) Concentrations
Description: Anti-glycoprotein E (gE) Ab concentrations were determined by Enzyme-Linked Immunosorbent Assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in micro international units per milliliter (mIU/mL).
Time Frame: At Month 108 post first dose of initial vaccination course in study Zoster-003 (NCT00434577).
Population: The analysis for persistence at month 108 was performed on the According-to-protocol (ATP) cohort analysis of immunogenicity at Year 9, which included subjects who complied with the protocol criteria and had immunogenicity results available up to the timepoint considered.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 68
mIU/mL | 9122.9 [7775.2 to 10704.1]

2. Primary Outcome: Anti-glycoprotein (gE) Specific Antibody (Ab) Concentrations
Description: Anti-gE Ab concentrations were determined by ELISA, presented as GMCs and expressed in mIU/mL.
Time Frame: At Month 120 post first dose of initial vaccination course in study Zoster-003 (NCT00434577).
Population: The analysis for persistence at month 120 was performed on the ATP cohort analysis of immunogenicity at Year 10, which included subjects who complied with the protocol criteria and had immunogenicity results available up to the timepoint considered.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 61
mIU/mL | 7384.0 [6202.8 to 8790.1]

3. Primary Outcome: Frequencies of gE (Glycoprotein)-Specific Cluster of Differentiation (CD4) (2+) T-cells.
Description: gE specific CD4 (2+) T-cells expressing at least 2 activation markers among IFN-γ, IL-2, TNF-α and CD40L, were determined by means of Intracellular Cytokine Staining (ICS) and expressed in T-cells/million cells.
Time Frame: At Month 108 post first dose of initial vaccination course in study Zoster-003 (NCT00434577).
Population: The analysis for persistence at month 108 was performed on the ATP cohort analysis of immunogenicity at Year 9, which included subjects who complied with the protocol criteria and had immunogenicity results available up to the timepoint considered.
Measure: Median (Inter-Quartile Range); unit: CD4 T-cells/million cells
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 66
CD4 T-cells/million cells | 414.0 [220.9 to 796.5]

4. Primary Outcome: Frequencies of gE (Glycoprotein)-Specific Cluster of Differentiation (CD4) (2+) T-cells.
Description: gE specific CD4 (2+)T-cells expressing at least 2 activation markers among IFN-γ, IL-2, TNF-α and CD40L were determined by means of ICS and expressed in T-cells/million cells.
Time Frame: At Month 120 post first dose of initial vaccination course in study Zoster-003 (NCT00434577).
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: CD4 T-cells/million cells
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 57
CD4 T-cells/million cells | 401.9 [298.1 to 901.9]

5. Secondary Outcome: Anti-glycoprotein (gE) Specific Antibody (Ab) Concentrations by Each Age Category
Description: Anti-gE Ab concentrations as determined by ELISA by each age category (60-69 years of age [YOA] and ≥70 YOA at the time of initial vaccination).Antibody concentrations were presented as GMCs and expressed in mIU/mL.
Time Frame: At Months 108 and 120 post first dose of initial vaccination course in study Zoster-003 (NCT00434577).
Population: The analysis for persistence at month 108 and 120 was performed on the ATP cohort analysis of immunogenicity at Years 9 and 10, which included subjects who complied with the protocol criteria and had immunogenicity results available at the time points considered.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Groups:
- GSK1437173A Vaccine 60-69 YOA Sub-group: Subjects of 60-69 YOA at the time of initial vaccination, who completed vaccination course of 2 doses of HZ/su vaccine (50 µg) in Zoster-003 (NCT00434577) study.
- GSK1437173A Vaccine ≥ 70 YOA Sub-group: Subjects aged 70 or more than 70 YOA at the time of initial vaccination, who completed vaccination course of 2 doses of HZ/su vaccine (50 µg) in Zoster-003 (NCT00434577) study.
Arm/Group | GSK1437173A Vaccine 60-69 YOA Sub-group | GSK1437173A Vaccine ≥ 70 YOA Sub-group
Number analyzed (Participants) | 13 | 55
mIU/mL
  Anti-gE, Month 108 | 8566.4 [5697.1 to 12880.9] | 9259.6 [7741.6 to 11075.2]
  Anti-gE, Month 120: number analyzed (Participants) | 11 | 50
  Anti-gE, Month 120 | 7401.4 [4894.2 to 11193.1] | 7380.2 [6048.9 to 9004.4]

6. Secondary Outcome: Frequencies of Antigen-specific CD4 (2+) T-cells by Each Age Category
Description: Antigen specific CD4 (2+) T-cells as determined by means of ICS and expressed in T-cells/million cells, by each age category (60-69 YOA and ≥ 70 YOA at the time of initial vaccination).
Time Frame: At Months 108 and 120 post first dose of initial vaccination course in study Zoster-003 (NCT00434577).
Population: The analysis for persistence at month 108 and 120 was performed on the ATP cohort analysis of immunogenicity at Years 9 and 10, which included subjects who complied with the protocol criteria and had immunogenicity results available at the timepoints considered.
Measure: Median (Inter-Quartile Range); unit: CD4 T-cells/million cells
Arm/Group | GSK1437173A Vaccine 60-69 YOA Sub-group | GSK1437173A Vaccine ≥ 70 YOA Sub-group
Number analyzed (Participants) | 13 | 53
CD4 T-cells/million cells
  CD4(2+), Month 108 | 453.8 [233.2 to 577.6] | 398.9 [220.9 to 811.3]
  CD4(2+), Month 120: number analyzed (Participants) | 11 | 46
  CD4(2+), Month 120 | 359.2 [254.9 to 885.0] | 429.4 [298.1 to 940.1]

7. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) Related to Study Participation or to a Concurrent GSK Medication/Vaccine (Including GSK1437173A Administered During the Zoster-003 [NCT00434577] Study).
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Between Months 108 and 120 post first dose of initial vaccination course in study Zoster-003 (NCT00434577).
Population: The analysis was performed on the Total enrolled cohort which included all subjects enrolled into the current study [ZOSTER-060 (NCT02735915)].
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 70
Participants | 0

8. Secondary Outcome: Anti-gE Specific Antibody (Ab) Concentrations
Description: Anti-gE antibody concentrations were determined by ELISA in all subjects, presented as GMCs and expressed in mIU/mL.
Time Frame: At 1 month post each re-vaccination dose (i.e. Month 121 and Month 123) and at 1 year post last re-vaccination dose (i.e., Month 134).
Population: The analysis was performed on the ATP cohort analysis of immunogenicity after re-vaccination, which included subjects who complied with the protocol criteria, have received at least one dose from the re-vaccination schedule and had immunogenicity results available at the timepoints considered.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 54
mIU/mL
  Anti-gE, Month 121 | 108199.6 [87154.2 to 134326.8]
  Anti-gE, Month 123 | 90003.6 [76754.3 to 105539.9]
  Anti-gE, Month 134: number analyzed (Participants) | 52
  Anti-gE, Month 134 | 30066.2 [25810.3 to 35023.8]

9. Secondary Outcome: Frequencies of Antigen-specific CD4 (2+) T-cells, Post Re-vaccination Course.
Description: Antigen specific CD4 (2+)T cells were determined by means of ICS and expressed in T-cells/million cells.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: CD4 T-cells/million cells
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 50
CD4 T-cells/million cells
  CD4(2+), Month 121: number analyzed (Participants) | 48
  CD4(2+), Month 121 | 2563.9 [1219.9 to 4127.4]
  CD4(2+), Month 123 | 1775.5 [1181.4 to 3077.8]
  CD4(2+), Month 134: number analyzed (Participants) | 48
  CD4(2+), Month 134 | 1196.3 [680.8 to 1850.8]

10. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms.
Description: Assessed solicited local symptoms included: pain, redness and swelling at injection site. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = significant pain at rest, prevented normal every day activities. Grade 3 redness/swelling = symptoms spreading beyond a surface of (>) 100 millimeters (mm).
Time Frame: Within 7 days (Days 0-6) after each vaccination and across doses, in the current study.
Population: The analysis was performed on the Total vaccinated cohort for re-vaccination course, which included all subjects with at least one dose of GSK1437173A vaccine in the current ZOSTER-060 (NCT02735915) study, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 62
Participants
  Any Pain, Dose 1 | 41
  Grade 3 Pain, Dose 1 | 1
  Any Redness, Dose 1 | 19
  >100 mm Redness, Dose 1 | 0
  Any Swelling, Dose 1 | 11
  >100 mm Swelling, Dose 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 56
  Any Pain, Dose 2 | 26
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 56
  Grade 3 Pain, Dose 2 | 2
  Any Redness, Dose 2: number analyzed (Participants) | 56
  Any Redness, Dose 2 | 17
  >100 mm Redness, Dose 2: number analyzed (Participants) | 56
  >100 mm Redness, Dose 2 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 56
  Any Swelling, Dose 2 | 7
  >100 mm Swelling, Dose 2: number analyzed (Participants) | 56
  >100 mm Swelling, Dose 2 | 0
  Any Pain, Across doses | 46
  Grade 3 Pain, Across doses | 2
  Any Redness, Across doses | 27
  >100 mm Redness, Across doses | 0
  Any Swelling, Across doses | 16
  > 100 mm Swelling, Across doses | 0

11. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms included: fatigue, gastrointestinal symptoms [nausea, vomiting, diarrhoea and/or abdominal pain], headache, myalgia, shivering and temperature [higher than or equal to (≥) 37.5 degrees Celsius (°C) for axillary, oral or tympanic route] and ≥38.0°C for rectal route. Grade 3 fatigue, gastrointestinal symptoms, headache, myalgia, shivering = symptoms that prevented normal activity. Grade 3 temperature = defined as fever higher than (>) 39.0°C, regardless of the route used.
Time Frame: Within 7 days (Days 0-6) after each vaccination and across doses, in the current study.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 62
Participants
  Any Fatigue, Dose 1 | 25
  Grade 3 Fatigue, Dose 1 | 3
  Related Fatigue, Dose 1 | 25
  Any Gastrointestinal symptoms, Dose 1 | 7
  Grade 3 Gastrointestinal symptoms, Dose 1 | 0
  Related Gastrointestinal symptoms, Dose 1 | 7
  Any Headache, Dose 1 | 12
  Grade 3 Headache, Dose 1 | 3
  Related Headache, Dose 1 | 12
  Any Myalgia, Dose 1 | 20
  Grade 3 Myalgia, Dose 1 | 1
  Related Myalgia, Dose 1 | 19
  Any Shivering, Dose 1 | 12
  Grade 3 Shivering, Dose 1 | 2
  Related Shivering, Dose 1 | 12
  Any Temperature, Dose 1 | 9
  >39.0°C Temperature, Dose 1 | 0
  Related Temperature, Dose 1 | 8
  Any Fatigue, Dose 2: number analyzed (Participants) | 56
  Any Fatigue, Dose 2 | 15
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 56
  Grade 3 Fatigue, Dose 2 | 1
  Related Fatigue, Dose 2: number analyzed (Participants) | 56
  Related Fatigue, Dose 2 | 14
  Any Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 56
  Any Gastrointestinal symptoms, Dose 2 | 7
  Grade 3 Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 56
  Grade 3 Gastrointestinal symptoms, Dose 2 | 0
  Related Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 56
  Related Gastrointestinal symptoms, Dose 2 | 5
  Any Headache, Dose 2: number analyzed (Participants) | 56
  Any Headache, Dose 2 | 12
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 56
  Grade 3 Headache, Dose 2 | 1
  Related Headache, Dose 2: number analyzed (Participants) | 56
  Related Headache, Dose 2 | 12
  Any Myalgia, Dose 2: number analyzed (Participants) | 56
  Any Myalgia, Dose 2 | 15
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 56
  Grade 3 Myalgia, Dose 2 | 2
  Related Myalgia, Dose 2: number analyzed (Participants) | 56
  Related Myalgia, Dose 2 | 14
  Any Shivering, Dose 2: number analyzed (Participants) | 56
  Any Shivering, Dose 2 | 8
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 56
  Grade 3 Shivering, Dose 2 | 2
  Related Shivering, Dose 2: number analyzed (Participants) | 56
  Related Shivering, Dose 2 | 8
  Any Temperature, Dose 2: number analyzed (Participants) | 56
  Any Temperature, Dose 2 | 8
  >39.0°C Temperature, Dose 2: number analyzed (Participants) | 56
  >39.0°C Temperature, Dose 2 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 56
  Related Temperature, Dose 2 | 7
  Any Fatigue, Across doses | 31
  Grade 3 Fatigue, Across doses | 3
  Related Fatigue, Across doses | 31
  Any Gastrointestinal symptoms, Across doses | 11
  Grade 3 Gastrointestinal symptoms, Across doses | 0
  Related Gastrointestinal symptoms, Across doses | 10
  Any Headache, Across doses | 18
  Grade 3 Headache, Across doses | 4
  Related Headache, Across doses | 18
  Any Myalgia, Across doses | 29
  Grade 3 Myalgia, Across doses | 3
  Related Myalgia, Across doses | 27
  Any Shivering, Across doses | 16
  Grade 3 Shivering, Across doses | 4
  Related Shivering, Across doses | 16
  Any Temperature, Across doses | 15
  >39.0°C Temperature, Across doses | 0
  Related Temperature, Across doses | 13

12. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs) According to the Medical Dictionary for Regulatory Activities (MedDRA) Classification in All Subjects.
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 30 days (Days 0-29) after each vaccination in the current study.
Population: The analysis was performed on the Total vaccinated cohort for re-vaccination course, which included all subjects with at least one dose of GSK1437173A vaccine in the current ZOSTER-060 (NCT02735915) study.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 62
Participants
  Any AEs | 14
  Any Grade 3 AEs | 1
  Any Related AEs | 5

13. Secondary Outcome: Number of Subjects With Any, Related and Fatal SAEs.
Description: SAEs assessed include medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: From Dose 1 of re-vaccination (Month 120) until study end (Month 134).
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 62
Participants
  Any SAEs | 7
  Related SAEs | 0
  Any Fatal SAEs | 0

14. Secondary Outcome: Number of Subjects With Any and Related Potential Immune-mediated Diseases (pIMDs).
Description: pIMDs assessed includes AEs that were autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Related pIMDs= pIMDs assessed by the investigator as related to the vaccination.
Time Frame: From Dose 1 of re-vaccination (Month 120) until study end (Month 134).
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Vaccine Group
Number analyzed (Participants) | 62
Participants
  Any pIMDs | 0
  Related pIMDs | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: During the 7 day (Day 0-6) post vaccination. Unsolicited symptoms: during the 30-day (Days 0-29) post-vaccination period; SAEs: From study start (Month 108) up to study end (Month 134).
Description: Reported adverse events data correspond to the total vaccinated cohort for revaccination phase
Arm/Group | GSK1437173A Vaccine Group
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 7/62
Other Adverse Events (participants affected / at risk) | 53/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Vaccine Group (N=62)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (2)
Septic shock (Infections and infestations) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Vaccine Group (N=62)
Gastrointestinal disorder (Gastrointestinal disorders) | 11 (14)
Nausea (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 16 (20)
Fatigue (General disorders) | 31 (40)
Injection site pruritus (General disorders) | 1 (1)
Pain (General disorders) | 46 (67)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 15 (17)
Swelling (General disorders) | 16 (18)
Cystitis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 29 (35)
Headache (Nervous system disorders) | 18 (24)
Erythema (Skin and subcutaneous tissue disorders) | 27 (36)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT02735915/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT02735915/SAP_001.pdf